CLINICAL TRIAL: NCT03824119
Title: Effect of Non-steroidal Anti-inflammatory Use on Blood Pressure in Women With Hypertensive Disorders of Pregnancy: A Randomized Open Label Trial
Brief Title: Postpartum NSAIDS and Maternal Hypertension
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Richard H. Lee, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-17-00959
Record Dates: First submitted 2019-01-04; First posted 2019-01-31 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Preeclampsia; Gestational Hypertension; Superimposed Preeclampsia; Chronic Hypertension in Obstetric Context
MeSH Terms: conditions — Pre-Eclampsia; Hypertension, Pregnancy-Induced | interventions — Ibuprofen; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Postpartum Care (Active Comparator): Subjects will receive NSAIDs (e.g. ibuprofen, ketorolac) for routine postpartum pain management.
  Interventions: Drug: Ibuprofen 600 mg
- Standard Postpartum Care without NSAIDs (Active Comparator): Subjects will receive standard postpartum care without NSAID administration for pain management. Acetaminophen or narcotics will be substituted for ibuprofen as indicated by provider.
  Interventions: Other: Standard Postpartum Care without NSAIDs

INTERVENTIONS:
Drug: Ibuprofen 600 mg — Standard postpartum care (including administration of NSAIDs)
  Other Names: Standard Postpartum Care
  Arms: Standard Postpartum Care
Other: Standard Postpartum Care without NSAIDs — NSAID administration will be withheld from this group.
  Arms: Standard Postpartum Care without NSAIDs

SUMMARY:
Previous studies have suggested that NSAID use causes an increase in blood pressure. Further, blood pressure elevation has been noted in women with pregnancy related hypertensive disease during the postpartum period. NSAIDs remain part of standard postpartum care in women with hypertensive disease. The objective of this study is to determine whether postpartum standard care withholding NSAID use is associated with a clinically significant reduction in postpartum hypertension in women with pregnancy induced hypertension. The investigators hypothesize that women with pregnancy induced hypertensive disease will be half as likely to have blood pressure elevation of 150/100 mmHg in the first 24 hours postpartum.

This study is an open label randomized trial of women with antepartum hypertension. Women will be randomized to receive standard postpartum care or standard postpartum care without NSAIDs. Blood pressure measurements and patient outcomes will be recorded. The study period will begin at the time of delivery and will end at the time of hospital discharge.

DETAILED DESCRIPTION:
The objective of this study is to determine whether the withholding of NSAID use is associated with a clinically significant decrease in postpartum hypertension in women with antepartum hypertension. The investigators are interested in whether the use of NSAIDs elevates blood pressure to greater than or equal to 150/100 mmHg (by either systolic or diastolic parameters) more frequently in hypertensive women. The investigators hypothesize that among participants with hypertensive disease associated with pregnancy, those who have NSAIDs withheld from standard postpartum care (experimental arm) will be half as likely to have an increase of blood pressure of 150/100 mmHg in the first 24 hours postpartum compared to participants receiving standard care that includes NSAIDs (control arm).

This trial is a randomized, open label study investigating the effect of NSAID use on blood pressure during the immediate postpartum period in women with chronic hypertension (cHTN) or pregnancy induced hypertension (PIH). The experimental group in this study will be women randomized to withholding NSAIDs during the study period, as women with hypertension routinely receive NSAIDs postpartum. Women with a diagnosis of pregnancy induced hypertension [gestational hypertension (gHTN), preeclampsia, superimposed preeclampsia, ] or cHTN will be enrolled antepartum and will be separated into two groups by the route of delivery: vaginal vs. cesarean delivery. Participants in the control arm will be assigned to receive standard care, which includes NSAIDs (ketorolac, ibuprofen) and participants in the experimental arm will be assigned to receive standard care with NSAIDs withheld in the postpartum period for the duration of hospitalization. The intervention period will last approximately 2-4 days and will conclude at the time of hospital discharge.

Blood pressure measurements will be obtained and recorded routinely in the postpartum period until hospital discharge. More frequent measurements may be performed in the event of severe blood pressure elevations at the discretion of the provider and treating clinical team. Complete Blood Count (CBC) on postpartum Day 1 will be performed as part of standard care. Additional laboratory evaluations will be performed at the discretion of the provider. In addition to blood pressure measurement, pain scale scores will be recorded daily using a Numeric Pain Scale Score. Initiation of anti-hypertensive medication, severe hypertension (BP 160/110 mmHg), treatment with magnesium sulfate and adverse maternal outcomes (cerebrovascular accident, congestive heart failure, pulmonary edema, eclamptic seizure, death) will be documented and abstracted from the medical record.

A power calculation to estimate the appropriate number of subjects needed to detect a difference of 30% in the primary outcome, with an alpha level of 0.05 and 80% power demonstrates that approximately 100 subjects per group (50 in the experimental group and 50 in the control group) will be needed for each delivery route tested (vaginal and cesarean).

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years or older delivering at LAC/USC Hospital
* Delivery occurring at or after 20 weeks gestation
* Diagnosis of antenatal hypertensive disorder: gestational hypertension, preeclampsia without severe features, preeclampsia with severe features, superimposed preeclampsia, eclampsia, chronic hypertension

Exclusion Criteria:

* HELLP Syndrome
* Renal dysfunction (Serum Creatinine >1.1 in current pregnancy)
* Known liver disease
* Low platelet count (<50,000 during hospital admission)
* Known sensitivity or allergy to ibuprofen or acetaminophen
* Use of therapeutic doses of anticoagulation
* Postpartum hemorrhage requiring blood transfusion
* Neonate with platelet disorder or thrombocytopenia in breastfeeding mother

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-12-11 (Actual); Primary Completion 2022-12-11 (Estimated); Study Completion 2022-12-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with blood pressure elevation | 24 hours postpartum
  Incidence of Systolic Blood Pressure of 150 mmHg or Diastolic Blood Pressure of 100 mmHg or above

SECONDARY OUTCOMES:
Proportion of participants with blood pressure elevation | 48, 72 and 96 hours postpartum
  Incidence of Systolic Blood Pressure of 150 mmHg or Diastolic Blood Pressure of 100 mmHg or above
Number of participants with eclamptic Seizure | Through study completion, up to 6 weeks postpartum
  Documented occurrence of new onset generalized tonic-clonic seizure(s) or coma in a woman with preeclampsia
Number of participants with stroke | Through study completion, up to 6 weeks postpartum
  New onset neurologic deficit associated with neuroimaging (CT scan or MRI) evidence of brain infarction or bleeding
Initiation of anti-hypertensive medication | Randomization through hospital discharge, an average of 3-7 days
  Provider documentation of initiation of anti-hypertensive medication (e.g. nifedipine, labetalol)
Pain numerical rating scale (NRS) score | Randomization through hospital discharge, measured daily, an average of 3-7 days
  Numerical pain scale score 0-10; 0= no pain and 10=worst possible pain; total score reported
Number of participants with renal failure | Through study completion, up to 6 weeks postpartum
  Creatinine >1.1 or doubled
Number of participants with pulmonary edema | Through study completion, up to 6 weeks postpartum
  Evidence of lung infiltrates on chest radiograph or CT scan
Number of participants who die | From the date of randomization through date of death from any cause, assessed up to 6 weeks postpartum
Length of hospital stay | Through hospital discharge, an average of 3-7 days
  Number of days from delivery to hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lee, MD, Principal Investigator — University of Southern California
Locations (1):
- LA County Hospital/University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pope JE, Anderson JJ, Felson DT. A meta-analysis of the effects of nonsteroidal anti-inflammatory drugs on blood pressure. Arch Intern Med. 1993 Feb 22;153(4):477-84. PMID 8435027
- [Background] Johnson AG, Nguyen TV, Day RO. Do nonsteroidal anti-inflammatory drugs affect blood pressure? A meta-analysis. Ann Intern Med. 1994 Aug 15;121(4):289-300. doi: 10.7326/0003-4819-121-4-199408150-00011. PMID 8037411
- [Background] Curhan GC, Willett WC, Rosner B, Stampfer MJ. Frequency of analgesic use and risk of hypertension in younger women. Arch Intern Med. 2002 Oct 28;162(19):2204-8. doi: 10.1001/archinte.162.19.2204. PMID 12390063
- [Background] Makris A, Thornton C, Hennessy A. Postpartum hypertension and nonsteroidal analgesia. Am J Obstet Gynecol. 2004 Feb;190(2):577-8. doi: 10.1016/j.ajog.2003.08.030. PMID 14981414
- [Background] Schoenfeld A, Freedman S, Hod M, Ovadia Y. Antagonism of antihypertensive drug therapy in pregnancy by indomethacin? Am J Obstet Gynecol. 1989 Nov;161(5):1204-5. doi: 10.1016/0002-9378(89)90666-2. PMID 2589441
- [Background] Wasden SW, Ragsdale ES, Chasen ST, Skupski DW. Impact of non-steroidal anti-inflammatory drugs on hypertensive disorders of pregnancy. Pregnancy Hypertens. 2014 Oct;4(4):259-63. doi: 10.1016/j.preghy.2014.06.001. Epub 2014 Jul 11. PMID 26104814
- [Background] Viteri OA, England JA, Alrais MA, Lash KA, Villegas MI, Ashimi Balogun OA, Chauhan SP, Sibai BM. Association of Nonsteroidal Antiinflammatory Drugs and Postpartum Hypertension in Women With Preeclampsia With Severe Features. Obstet Gynecol. 2017 Oct;130(4):830-835. doi: 10.1097/AOG.0000000000002247. PMID 28885417
- [Background] Vigil-De Gracia P, Solis V, Ortega N. Ibuprofen versus acetaminophen as a post-partum analgesic for women with severe pre-eclampsia: randomized clinical study. J Matern Fetal Neonatal Med. 2017 Jun;30(11):1279-1282. doi: 10.1080/14767058.2016.1210599. Epub 2016 Aug 2. PMID 27384376
- [Background] Walters BN, Thompson ME, Lee A, de Swiet M. Blood pressure in the puerperium. Clin Sci (Lond). 1986 Nov;71(5):589-94. doi: 10.1042/cs0710589. PMID 3769407
- [Background] Hypertension in pregnancy. Report of the American College of Obstetricians and Gynecologists' Task Force on Hypertension in Pregnancy. Obstet Gynecol. 2013 Nov;122(5):1122-1131. doi: 10.1097/01.AOG.0000437382.03963.88. No abstract available. PMID 24150027
- [Background] Sibai BM. Etiology and management of postpartum hypertension-preeclampsia. Am J Obstet Gynecol. 2012 Jun;206(6):470-5. doi: 10.1016/j.ajog.2011.09.002. Epub 2011 Sep 16. PMID 21963308